CLINICAL TRIAL: NCT01337856
Title: Efficacy of Alcohol Hand-rubbing Covering All Hand Surfaces in Reducing Bacterial Hand Contamination of Healthcare Staff
Acronym: B/07/310
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Angela Chow, Tan Tock Seng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NHG DSRB B/07/310; SIG08012 (Other Grant/Funding Number: National Healthcare Group)
Record Dates: First submitted 2011-04-13; First posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Efficacy of Hand Hygiene Protocols
Keywords: time-effectiveness; hand hygiene protocols
MeSH Terms: interventions — Hand Hygiene; Ethanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- WHO alcohol handrub protocol (Other): handrubbing with alcohol using the standard 7-step technique (WHO alcohol handrub protocol)
  Interventions: Other: Hand hygiene protocol
- CDC alcohol handrub protocol (Other): Handrubbing with alcohol covering all hand surfaces in no particular order (CDC alcohol handrub protocol)
  Interventions: Other: Hand hygiene protocol
- Chlorhexidine handwashing (Other): chlorhexidine handwashing using the standard 7-step technique (WHO handwashing protocol)
  Interventions: Other: Hand hygiene protocol

INTERVENTIONS:
Other: Hand hygiene protocol — Comparison of efficacy of 3 hand hygiene protocols
  Other Names: time-effectiveness; efficacy; hand hygiene; alcohol handrub

SUMMARY:
This is a randomized controlled trial comparing the effectiveness of three hand hygiene protocols, during routine inpatient clinical care: Protocol 1: handrubbing with alcohol covering all hand surfaces in no particular order; Protocol 2: handrubbing with alcohol using the WHO standard 7-step technique; and Protocol 3: handwashing with chlorhexidine using the WHO standard 7-step technique.

The main study hypothesis is that alcohol hand-rubbing covering all hand surfaces is not less effective in reducing bacterial hand contamination of healthcare staff than alcohol hand-rubbing using 7-step technique; and is more effective than chlorhexidine handwashing. The secondary study hypothesis is that time spent on alcohol hand-rubbing covering all hand surfaces is less than that required by the other 2 hand hygiene protocols respectively.

DETAILED DESCRIPTION:
Background

1. The hospital environment is conducive for the rapid spread of pathogens, especially antimicrobial-resistant bacteria. Hospital-acquired methicillin-resistant staphylococcus aureus (MRSA) and vancomycin-resistant enterococci (VRE) infections are increasing worldwide, including Singapore.
2. Good hand hygiene is the single most important measure to prevent the nosocomial spread of pathogens in healthcare settings. However, most studies have reported compliance rates of <50%, under routine hospital practice. The last hand hygiene audit in TTSH revealed a compliance rate of merely 20%. Recent studies have observed that this level of compliance would not reduce the transmission risk of multi-resistant bacteria in the hospital. A high workload and insufficient time for hand hygiene are common reasons cited by healthcare workers for poor compliance with hand hygiene.
3. Hospital staff are responsible for 20-40% of nosocomial spread of pathogens from patient to patient through contact transmission. Bacterial contamination of healthcare workers' hands during routine patient care has been reported to increase linearly with time, with an average increase of 16 colony-forming units (CFUs) per minute of patient care.
4. The use of alcohol handrubs has been demonstrated to significantly reduce time spent on hand hygiene (40-80 seconds required for hand-washing vs 20 seconds for alcohol hand-rubbing). Although there is growing evidence from experimental studies that alcohol-based products are more effective than soap or antimicrobial soaps, there have been very few trials done in the clinical setting evaluating the two hand hygiene protocols in everyday practice.
5. A randomised controlled trial carried out in 3 intensive care units (ICUs) of a 940-bedded French tertiary care and referral university hospital demonstrated the superior antimicrobial efficacy of alcohol hand-rubbing compared with chlorhexidine hand-washing. The median percentage reduction in bacterial contamination was significantly higher with alcohol hand-rubbing than with hand-washing (83% vs 58%, p = 0.012). Another randomised clinical trial involving 4 general wards and 3 ICUs at the 850-bedded University of Barcelona Hospital demonstrated similar findings. It reported an average reduction in hand bacterial load of 88.2% with alcoholic hand-wash, compared with 49.6% with regular liquid soap.
6. Since the introduction of alcohol handrubs at Tan Tock Seng Hospital (TTSH), the hospital has adopted the hand hygiene guidelines issued by the Centers for Disease Control and Prevention (CDC). The CDC guidelines do not specifically discuss the technique for using alcohol-based handrubs. However, the recent World Health Organization (WHO)'s Guidelines on Hand Hygiene in Health Care (Advanced Draft) April 2006 have detailed the hand hygiene technique with alcohol-based formulation. WHO's recommended alcohol hand-rubbing technique involves the same standard 7-steps adopted in hand-washing with antiseptic soap and water.
7. Busy healthcare staff are often unable to adhere to the 7-step hand hygiene technique. Hence, the most convenient hand hygiene protocol would be hand-rubbing with alcohol, covering all hand surfaces until dry, as recommended by the CDC. This is the protocol currently adopted by TTSH. However, there has been growing concern that there could be missed areas on the hands after alcohol hand-rubbing, which might affect the efficacy of the alcohol handrub [20, 21].
8. There have been very few published clinical studies comparing the efficacy of alcohol hand-rubbing with antiseptic hand-washing in healthcare workers during routine patient care. To our knowledge, there has not been a published international study comparing CDC's recommended alcohol hand-rubbing protocol with that of the WHO's. This study will provide important information on the efficacy of alcohol hand-rubbing using the current technique adopted in TTSH (CDC's guidelines), compared with the WHO's recommended 7-step technique for alcohol hand-rubbing and the standard 7-step chlorhexidine hand-washing respectively. This study will also provide local data on the actual time spent on hand hygiene, during everyday practice. The findings from this study will contribute significantly towards understanding hand hygiene practices during routine patient care in our local healthcare setting and hence guide infection control strategies to reduce hospital-acquired infections. Reducing hospital-acquired infections would lead to improved clinical outcomes for our patients.

   Study Hypothesis:
9. Alcohol hand-rubbing covering all hand surfaces is not less effective in reducing bacterial hand contamination of healthcare staff than alcohol hand-rubbing using 7-step technique; and is more effective than chlohexidine handwashing. Time spent on alcohol hand-rubbing covering all hand surfaces is less than that required by the other 2 hand hygiene protocols respectively.

   Objectives
10. The primary objective of this study is to evaluate the efficacy of 3 hand hygiene protocols: hand-rubbing with alcohol covering all hand surfaces, hand-rubbing with alcohol using the standard 7-step technique, and hand-washing with chlorhexidine using the standard 7-step technique. The secondary objectives include the estimation of time spent on hand hygiene, for each hand hygiene protocol; and the evaluation of bacterial hand contamination after key patient care activities.

    Methods
11. This study will be a prospective randomised controlled trial, with blinded evaluation of microbiological results. Three hand hygiene protocols will be compared: hand-rubbing with alcohol covering all hand surfaces, hand-rubbing with alcohol using the standard 7-step technique, and hand-washing with chlorhexidine using the standard 7-step technique.
12. Medical and nursing staff from general wards in TTSH will be invited to participate in the study. 60 medical staff (namely medical officers and house officers) and 60 nursing staff (namely registered nurses and enrolled nurses) will be recruited for the study. The medical and nursing teams working in the selected wards will be informed of the study prior to its commencement, and the support of the respective unit and department heads sought. An information sheet describing the study will be circulated prior to the study.
13. The study will be carried out over 8 weeks, during the day shifts, from Monday to Friday. Two infection control nurses and a research associate will work as a team, moving systematically from one ward to the next. On the day of the study, the team will observe the patient care activities in the participating ward, and look out for activities involving direct patient contact (such as physical examination, temperature or blood pressure taking), without the use of gloves.
14. Whenever a medical or nursing staff is about to perform an activity involving direct patient contact without the use of gloves, the staff will be approached and invited to participate in the study. Verbal consent will be taken from staff who accept the invitation to participate. To protect the identity and confidentiality of the participating staff, written consent will not be taken.
15. Three samples for bacterial counts will be taken from the dominant hand of each participant: just prior to patient contact, after patient contact, and after hand hygiene.
16. Each participant will be randomly assigned to one of the 3 hand hygiene protocols:

    * hand-rubbing with alcohol covering all hand surfaces,
    * hand-rubbing with alcohol using the standard 7-step technique, or
    * hand-washing with chlorhexidine using the standard 7-step technique. Pre-prepared sealed envelopes will be used. Participants allocated into hand hygiene protocols (1) and (3) will be asked to perform the hand hygiene method, as they normally would. Participants assigned to hand hygiene protocol (2) will be requested to perform hand-rubbing with alcohol, using the technique they would normally adopt for chlorhexidine hand-washing.
17. The two infection control nurses will separately monitor the time taken by each participant for the patient care activity using a stopwatch, and record the duration and type of patient care performed in the data collection form. The data collection form will only contain a study number and will not bear the name or identification of the participant. A study number will be randomly assigned to each participant using pre-numbered data collection forms. Similarly, the infection control nurses will observe and record the duration of each hand hygiene and note adherence to the allocated hand hygiene technique. The infection control nurses will only make observations, and will not interfere with hand hygiene whatever the method used. (Pls see attached data collection form)
18. Participants assigned to one of the 2 alcohol hand-rubbing protocols but whose hands become visibly soiled after patient care, will be advised to perform chlorhexidine hand-washing instead.
19. The research associate, who has undergone training in the sampling technique, will be responsible for taking hand samples for bacterial counts, using the glove juice technique. Samples will be labelled with study numbers only. Innoculated agar plates will be incubated at 37 degC under aerobic conditions. The total bacterial contamination of hands in terms of the number of colony forming units (cfu) will be recorded after 48 hours of incubation. Bacteria present in the samples will also be qualitatively identified and reported. The microbiologist examining the culture plates and reporting the microbiological results will be blinded to the hand hygiene method used.
20. Each staff will only be approached once. The time taken for each sample collection will be less than a minute. The study team will ensure that the study will not interfere with routine patient care activities.
21. Strict confidentiality of participants will be maintained. All data collected, including microbiological results, will be identified only by the study number and cannot be traced to the participating staff.

ELIGIBILITY:
Inclusion Criteria:

medical and nursing staff working in general wards in Tan Tock Seng Hospital

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
reduction of hand bacterial load | hand samples will be analyzed up to 11 months after collection; data will be presented for an average of 5 years after data collection
  The primary outcome measure of the study was to ascertain the effectiveness of the three hand-hygiene protocols, in the reduction of hand bacterial load. Quantitative reduction in bacterial load will be measured in colony forming units per mililiter (cfu/ml). Bacteria will be qualitatively identified, and sensitivity to antibiotics determined.

SECONDARY OUTCOMES:
time spent on hand hygiene | participants will be observed for the duration of hand hygiene; data will be presented for an average of 5 years after data collection
  The secondary outcome measure include the estimation of time spent on hand hygiene, for each hand hygiene protocol. Time will be measured in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Angela LP Chow, MBBS, MPH, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore, Singapore